CLINICAL TRIAL: NCT04812028
Title: Magnesium Sulfate as Adjuvant Analgesia and Its Effect on Opiate Use of Post-operative Transplant Patients in the Pediatric ICU
Brief Title: Magnesium Sulfate for Analgesia in Pediatric Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2019-27677
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prospective Experimental Group (Experimental): Participants in this group will prospectively receive the intervention.
  Interventions: Drug: Magnesium sulfate
- Retrospective Review Group (No Intervention): Participants in this group will have their medical records retrospectively reviewed.

INTERVENTIONS:
Drug: Magnesium sulfate — Magnesium sulfate (MgSO4) will be administered intravenously at induction of anesthesia as a 30-minute bolus dose of 50 mg/kg (maximum 2 grams) in the OR, followed by a 15 mg/kg/hr IV infusion for 48 hours or once the patient has transferred out of the PICU, whichever comes first.
  Arms: Prospective Experimental Group

SUMMARY:
To use magnesium sulfate as adjuvant analgesia by implementing a treatment protocol in order to determine whether can benefit pediatric pain in post-operative transplanted patients and decrease overall opioid consumption.

DETAILED DESCRIPTION:
The post-operative ICU course for children receiving liver transplants and TPIAT (total pancreatectomy with islet cell autotransplantation) includes a number of different challenges, one of which includes pain. Pain is treated with both medications and approaches without medications (such as music and other distraction techniques). Opioids are one such effective pain medication which is universally used, however like all medications has risks of certain side effects (such as nausea, constipation, itching, and others). Modern research has searched for other medications and methods to treat pain in both children and adults. In this study, the investigators aim to apply one of these methods that has been shown to be effective in certain operative populations through a medicine called Magnesium-Sulfate, which may be a safe way to decrease the use of other pain medications (specifically opioids). Magnesium is already a physiologic electrolyte the body uses, which are consumed from certain foods. Used as an IV medication to reach higher levels of magnesium can work to decrease pain via its action on specific nerve receptors. Magnesium-Sulfate will be given at the beginning of transplant surgery for consented liver and TPIAT transplant patients, and continue an infusion for 48 hours into their ICU course. The investigators will monitor side effects and treat pain the same way otherwise the care team would without magnesium to determine whether there is any beneficial effect that can be applied to children in the future.

ELIGIBILITY:
Inclusion Criteria:

Experimental Group:

- Be scheduled for and receive a liver transplant or total pancreatectomy and islet cell autotransplantation

Control Group:

- Received a liver transplant or total pancreatectomy and islet cell autotransplantation.

Exclusion Criteria:

Experimental Group:

* Pregnant or unwilling to abstain from sex if not practicing birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Known allergic reactions to components of the MgSO4
* History of heart block or myasthenia graves in past medical history.
* Presence of cardiac pacemaker
* Any patient with preoperative creatinine level > 1.5x upper limit of normal.

Control Group:

* Any patient who had filed as research-exempt (opt-out of research previously).
* Any patient with preoperative creatinine level > 1.5x upper limit of normal.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwenyth Fischer, MD, Principal Investigator — University of Minenesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Liver Transplant - MgSO4: Liver transplant recipients receiving study intervention (magnesium sulfate infusion)
- TPIAT - MgSO4: Total Pancreatecomy with Islet Cell Autotransplantation (TPIAT) recipients receiving study intervention (MgSO4 infusion)
- Liver Transplant - Control Review Group: Retrospective cohort of liver transplant recipients whom did not receive study intervention
- TPIAT - Control: Retrospective cohort of TPIAT recipients whom did not receive study intervention
Period: Overall Study
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Started | 2 | 9 | 21 | 34
Completed | 2 | 9 | 21 | 34
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control | Total
Number analyzed (Participants) | 2 | 9 | 21 | 34 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 9 | 21 | 34 | 66
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 9 | 21 | 38
  Male | 0 | 3 | 12 | 13 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 1 | 8 | 0 | 0 | 9
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 21 | 34 | 55

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Requirement
Description: Total opioid requirement during the entire operative and post-operative pediatric intensive care unit (PICU) period will be reported in units of morphine equivalent per body weight.
  OME/kg is often the recorded value in studies, however the patients had variable PICU courses (i.e. duration in days different between patients, as well as well as admission times altering POD#0 data, etc), so the opioid consumption was standardized to the duration of their course (i.e. OME/kg/d).
Time Frame: approximately 7 days
Measure: Mean (Standard Deviation); unit: OME/kg/d
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
OME/kg/d | 3.31 (1.69) | 5.27 (2.94) | 10.2 (8.32) | 4.1 (2.41)

2. Secondary Outcome: Daily Post-operative Opioid Requirement
Description: Daily opioid requirement will be reported in units of morphine equivalent per body weight.
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5
Measure: Mean (Standard Deviation); unit: OME/kg/d
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
OME/kg/d | 4.3 (1.28) | 5.33 (3.03) | 14.06 (11.6) | 4.97 (3.28)

3. Secondary Outcome: OR Opioid Consumption
Description: Oral Morphine Equivalent use during Operating Room Procedure
  OME/kg is often the recorded value in studies, however the patients had variable PICU courses (i.e. duration in days different between patients, as well as well as admission times altering POD#0 data, etc), so the opioid consumption was standardized to the duration of their course (i.e. OME/kg/d).
Time Frame: approximately 7 days
Measure: Mean (Standard Deviation); unit: OME/kg/d
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
OME/kg/d | 2.19 (0.3) | 3.6 (2.51) | 4.69 (1.94) | 3.24 (1.44)

4. Secondary Outcome: Opioid Side Effect - Delirium/AMS
Description: Outcome reported as the count of participants who experience opioid side effects during the entire operative and post-operative pediatric intensive care unit (PICU) period.
  Delirium or Altered Mental Status
Time Frame: approximately 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
Participants | 0 | 5 | 5 | 7

5. Secondary Outcome: Opioid Side Effect - Constipation -- Ileus
Description: Outcome reported as the count of participants who experience opioid side effects during the entire operative and post-operative pediatric intensive care unit (PICU) period.
  Prevalence of Ileus as indicated in Progress Note
Time Frame: approximately 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
Participants | 0 | 5 | 5 | 21

6. Secondary Outcome: Opioid Side Effect - Constipation -- Enema Use
Description: Outcome reported as the count of participants who experience opioid side effects during the entire operative and post-operative pediatric intensive care unit (PICU) period.
  Prevalence of enema use for constipation
Time Frame: approximately 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
Participants | 0 | 2 | 5 | 11

7. Secondary Outcome: Opioid Side Effect - Constipation -- 1st Stool
Description: Postoperative day where first stooled
Time Frame: approximately 7 days
Measure: Mean (Full Range); unit: day
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
day | 2 [1 to 3] | 4 [1 to 6] | 3.83 [0 to 7] | 3.76 [1 to 5]

8. Secondary Outcome: Opioid Side Effect - Bowel Dysmotility -- Feed Initiation
Description: Postoperative day where started enteral feeds
Time Frame: approximately 7 days
Measure: Mean (Full Range); unit: day
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
day | 2 [1 to 3] | 2.22 [1 to 4] | 2.71 [1 to 6] | 2.06 [1 to 4]

9. Secondary Outcome: Opioid Side Effect - Nausea -- Emeses
Description: Postoperative number of emeses as indicator of nausea
Time Frame: approximately 7 days
Measure: Mean (Full Range); unit: events
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
events | 0 [0 to 0] | 2.44 [0 to 9] | 1.38 [0 to 5] | 1.26 [0 to 6]

10. Secondary Outcome: Opioid Side Effect - Nausea -- Antiemetic Use
Description: Number of ondansetron doses
Time Frame: approximately 7 days
Measure: Mean (Standard Deviation); unit: antiemetic administrations
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
antiemetic administrations | 1 (1.41) | 11.4 (11.95) | 2.86 (4.65) | 10.79 (9.24)

11. Secondary Outcome: Opioid Side Effect - Nausea -- Antiemetic Use
Description: Frequency needing any antiemetic use, measure reported in percentage
Time Frame: approximately 7 days
Measure: Number; unit: percentage
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
percentage | 50 | 89 | 43 | 94

12. Secondary Outcome: Opioid Side Effect - Pruritus
Description: Frequency of pruritus as measured by Naloxone gtt use, reported as percentage
Time Frame: approximately 7 days
Measure: Number; unit: percentage
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
percentage | 0 | 78 | 14 | 59

13. Secondary Outcome: Opioid Side Effect - Urinary Retention
Description: Frequency of urinary retention as measured by straight catheterization requirement, measured in percentage
Time Frame: approximately 7 days
Measure: Number; unit: percentage
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
percentage | 0 | 22 | 10 | 18

14. Secondary Outcome: PICU Length of Stay
Description: Consecutive days in PICU following operation
Time Frame: up to 32 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Liver Transplant - MgSO4 | TPIAT - MgSO4 | Liver Transplant - Control Review Group | TPIAT - Control
Number analyzed (Participants) | 2 | 9 | 21 | 34
days | 4.19 (0.42) | 7.38 (2.92) | 8.47 (6.97) | 7.29 (7.67)

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- Liver Transplant - MgSO4 Group: Liver transplant recipients receiving study intervention (magnesium sulfate infusion)
- Liver Transplant - Control: Retrospective cohort of liver transplant recipients whom did not receive study intervention
Arm/Group | Liver Transplant - MgSO4 Group | TPIAT - MgSO4 | Liver Transplant - Control | TPIAT - Control
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/9 | 0/21 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/9 | 0/21 | 0/34
Other Adverse Events (participants affected / at risk) | 2/2 | 7/9 | 17/21 | 27/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liver Transplant - MgSO4 Group (N=2) | TPIAT - MgSO4 (N=9) | Liver Transplant - Control (N=21) | TPIAT - Control (N=34)
Hypotension (General disorders) | 2 | 7 | 17 | 27
Bradycardia (General disorders) | 0 | 3 | 13 | 8
Aryrthmia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2
Delirium/Hallucination (General disorders) | 0 (0) | 5 (5) | 4 (4) | 7 (7)
Pulmonary Edema/Efusion (General disorders) | 1 (1) | 2 (2) | 7 (7) | 2 (2)
Infecrion (General disorders) | 0 (0) | 4 (4) | 4 (4) | 15 (15)
Prolonged Hypoxia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anaphlaxis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
abnormal movement or sensation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
AKI (General disorders) | 1 (1) | 0 (0) | 7 (7) | 1 (1)
Flushing (General disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT04812028/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT04812028/ICF_001.pdf